CLINICAL TRIAL: NCT04005209
Title: Early Low-dose Ketamine Infusion Versus Usual Care for Sickle Cell Pain Crisis: a Randomized, Prospective Study.
Brief Title: Ketamine Infusion for Sickle Cell Pain Crisis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Decided not to open study
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100887
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Anemia; Sickle-Cell, With Crisis; Acute Pain
Keywords: Ketamine; Intravenous Infusions; Anemia; Sickle-Cell, with Crisis; Acute Pain
MeSH Terms: conditions — Vaso-Occlusive Crises; Acute Pain | interventions — Ketamine; Pain Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pain management without ketamine infusion (Active Comparator): Pain management without ketamine infusion. No other restrictions on pain management or medications.
  Interventions: Other: Pain management
- Pain management with ketamine infusion (Experimental): Pain management that includes a ketamine infusion. No other restrictions on pain management or medications.
  Interventions: Drug: Ketamine; Other: Pain management

INTERVENTIONS:
Drug: Ketamine — The experimental group will receive a ketamine intravenous infusion, initiated at 0.2 mg/kg/hr within the first 12 to 24 hours on an inpatient admission for sickle cell pain crisis, and titrated per hospital policy by the inpatient pain service.
  Arms: Pain management with ketamine infusion
Other: Pain management — Pain management

SUMMARY:
The purpose of this study is to prospectively study the efficacy of low dose ketamine infusions in treating patients who are admitted to the hospital with a sickle cell pain crisis. Participants will be prospectively randomized in unblinded fashion in the first 12 to 24 hours of an inpatient admission for sickle cell pain crisis to receive pain management without ketamine infusion (Group A) versus pain management that includes low-dose ketamine infusion starting at 0.2mg/kg/h (Group B). The effect of this intervention on various pain management and healthcare utilization outcome measures will be recorded and analyzed to determine whether or not there is a measurable benefit of using ketamine infusions in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Have a pre-existing/known diagnosis of sickle cell disease, prior to the current presentation
* Admitted to Duke University Hospital with a clinical diagnosis of sickle cell crisis
* Are at least 18 years old at time of admission
* Have been admitted to any hospital for sickle cell pain crisis at least twice in the last year
* Have documented severe pain at time of admission, requiring intravenous opiates
* Must be able to speak English

Exclusion Criteria:

* Are greater than 70 years old at time of admission
* Carry a diagnosis of cirrhosis, elevated intracranial pressure, elevated intraocular pressure, active coronary artery disease, and psychiatric disorders with history of psychosis
* Are pregnant or breastfeeding
* Are concomitantly admitted for another medical or surgical problem in addition to sickle cell pain crisis
* Have been admitted to any hospital for a sickle cell pain crisis greater than 10 times in the last year
* Were admitted to any hospital for sickle cell pain crisis within the last 30 days
* Are able to fully and properly consent for their own medical care, with no restrictions or limitations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in grand mean opioid consumption from 0 to 72 hours | baseline, 72 hours

SECONDARY OUTCOMES:
Percentage reduction in grand mean pain score using the 11-point visual analog scale | baseline, 72 hours
  Using standard 11-point visual analog pain scale, ranging from 0 = no pain to 10 = worst pain imaginable.
Time from inpatient admission to readiness for discharge | Upon discharge from the hospital (an average of 1 week)
30-day hospital readmission rate | 30 days from discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No